CLINICAL TRIAL: NCT06085287
Title: Electromagnetic Therapy for Autism Spectrum Disorder: a Pilot Randomized Controlled Trial
Brief Title: Electromagnetic Therapy for Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lo Kwai Ching, Assistant Lecturer, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 23-273
Record Dates: First submitted 2023-07-06; First posted 2023-10-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; ASD; EMT; Electromagnetic therapy; Chinese Medicine
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Magnetic Field Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAU+EMT groups (Experimental): CAU+EMT group will continue their current interventions and medications as usual. The existing interventions and medications will be recorded and serve as covariates included in outcome analysis. Besides, CAU+EMT group will receive a total of 30 sessions of EMT within 12 weeks (2 - 3 sessions/week).
  Interventions: Device: Electromagnetic therapy
- CAU Group (No Intervention): CAU group will continue their current interventions and medications as usual. The existing interventions and medications will be recorded and serve as covariates included in outcome analysis.Those who are initially assigned to CAU group will receive EMT for 12 weeks after they complete the trial. The post-trial treatment will serve as a compensation for their participation.

INTERVENTIONS:
Device: Electromagnetic therapy — Electromagnetic therapy will be performed using an electromagnetic stimulator (Smart Cap). Chinese medicine practitioners who have at least 3 years of experience will conduct EMT after training. Each session of EMT will take 20-25 min, with 2-3 sessions per week, total of 30 sessions finished within 12 weeks.
  Arms: CAU+EMT groups

SUMMARY:
The investigators hypothesize that electromagnetic therapy (EMT) could produce greater improvement on Autism spectrum disorder (ASD) compared to the waitlist control. To test this hypothesis, a pilot randomized waitlist-controlled trial is designed to achieve the 2 aims:

1. To evaluate the efficacy of EMT in improving children with ASD as measured by Childhood Autism Rating Scale (CARS) by comparing the change in CARS scores from baseline to week 12 between the two groups.
2. To assess the safety of EMT by comparing the number of participants with adverse events, number of participants withdrawn and reasons of withdrawal in treatment group with those in the control group.

A pilot randomized waitlist-controlled trial is designed. A total of 30 children aged 3-12 years with a principal diagnosis of ASD will be recruited. They will be randomly assigned to Care-As Usual (CAU) and CAU+EMT groups (n = 15 each group). Participants on the CAU+EMT group will receive a total of 30 sessions of EMT within 12 weeks (2 - 3 sessions/week).Those who are initially assigned to CAU group will receive EMT for 12 weeks after they complete the trial. The post-trial treatment will serve as a compensation for their participation.

ELIGIBILITY:
Inclusion Criteria:

1. aged 3-12 years;
2. have had a principal diagnosis of ASD according to the diagnostic criteria for ASD in the DSM-5;
3. The score of CARS is 30-37 (mild to moderate ASD) at entry; and
4. his/her parents or legal guardian give a written informed consent that indicates the permission to participate in the study.

Exclusion Criteria:

1. Children suffer a significant comorbid congenital disease or brain injury, such as Down syndrome, mental retardation, and cerebral palsy;
2. Children have been suffering uncontrolled epilepsy or seizure;
3. Children have heart diseases;
4. Children have participated in other investigational studies in previous 3 months;
5. Children have pediatric massage or acupuncture in previous 2 months; or
6. they have severe skin lesions or scar on the areas the treatment will be performed.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale（CARS） | The changes from baseline to week 12, week 24 and week 36.
  CARS consists of 15 items that cover all domains of ASD symptoms: 1, relationship to people; 2, Imitation; 3, emotional response; 4, body use; 5, object use; 6, adaptation to change; 7, visual response; 8, listening response; 9, taste-smell-touch response and use; 10, fear and nervousness; 11, verbal communication; 12. non-verbal communication; 13. Activity level; 14. Level and consistency of intellectual response; 15, general impressions. Each item is scored from "1" (normal behavior) to "4" (severely abnormal behavior), with a total score ranging from 15 to 60. Scores 30-37 indicate mild to moderate ASD; 38-60 indicate severe.

SECONDARY OUTCOMES:
Autism Treatment Evaluation Scale (ATEC) | The changes from baseline, week 12, week 24 and week 36.
  Autism Treatment Evaluation Scale is evaluated by a parent and serve as supplementary to CARS.The minimum vale of ATEC is 0 and the maximum value is 197, the higher the score the worse the outcome.
Children's Sleep Habits Questionnaire (CSHQ) | The changes from baseline, week 12, week 24 and week 36.
  The minimum vale of CSHQ is 0 and the maximum value is 66, the higher the score the worse the outcome.
Clinical Global Impression-Severity (CGI-S) | The changes from baseline, week 12, week 24 and week 36.
  The minimum vale of CGI-S is 0 and the maximum value is 7, the higher the score the worse the outcome.
Clinical Global Impression Severity-Improvement (CGI-I) | The changes from baseline, week 12, week 24 and week 36.
  The minimum vale of CGI-I is 0 and the maximum value is 7, the higher the score the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kwai Ching Lo, PHD, Principal Investigator — The University of Hong Kong
Locations (1):
- Clinical Services Centres, The School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes